CLINICAL TRIAL: NCT05095051
Title: A Novel Limb Cryocompression System for Prevention of Chemotherapy Induced Peripheral Neuropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Paxman Coolers Ltd. (Unknown); The N.1 Institute for Health, National University of Singapore (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 2021/00288
Record Dates: First submitted 2021-09-19; First posted 2021-10-27 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
Keywords: Chemotherapy-induced Peripheral Neuropathy; Cryocompression

STUDY DESIGN:
Intervention Model Description: Healthy subjects will undergo cryocompression of the various temperature and pressure levels in the cryocompression device. One temperature will be tested on 3 subjects for 3 hours. Tolerability of the temperature will be determined through a visual analogue pain scale (VAS). Should 1 out of 3 subjects display intolerance to the temperature level, 3 more healthy subjects will be tested to ensure consistency.
  Cancer patient limb cryocompression sessions will comprise of a pre-cooling period, continued with paclitaxel infusion and a post-cooling period. Overall, hypothermia will be administered for no longer than four hours.
  Each patient will undergo maximum limb cooling. The initial device settings for the first cycle for each patient will be based on the optimal temperature determined to be safe and tolerable in healthy subjects. Safety and tolerance of the concomitant cryocompression will be measured using VAS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy subjects (Experimental): To assess safety and tolerability of limb cryocompression, as well as to determine the optimal temperature and pressure to be used. The occurrence or lack of core hypothermia will be studied.
  Interventions: Device: Paxman Cryocompression System (PCCS)
- Cancer patients (Experimental): Once the optimal temperature and pressure of limb cryocompression is established in healthy subjects, a group of cancer patients will undergo limb cryocompression over multiple cycles of chemotherapy to establish safety and tolerability of repeated therapy.
  Interventions: Device: Paxman Cryocompression System (PCCS)

INTERVENTIONS:
Device: Paxman Cryocompression System (PCCS) — Establishing optimal temperature and pressure for limb cryocompression therapy. Healthy subjects will undergo 3 hours of limb cryocompression.
  The cryocompression device used in this study consists of a control unit, and limb wraps. The control unit contains the coolant reservoir and pump to circulate the coolant and air for compression. It is able to thermoregulate (control the temperature of the circulating coolant) and offer cyclic air pressure in the wraps. The wraps cover the limbs from the elbow/knee to the fingers/toes.
  Arms: Healthy subjects
Device: Paxman Cryocompression System (PCCS) — The study population will comprise of cancer patients scheduled to receive weekly paclitaxel chemotherapy for a maximum of 12 cycles.
  Paclitaxel will be administered as a one-hour infusion. Limb cryocompression sessions comprised of a pre-cooling period (up to one hour), continued with paclitaxel infusion and a post-cooling period (on average 30 minutes after the end of paclitaxel infusion). Overall, limb cryocompression will be administered for no longer than four hours.
  Arms: Cancer patients

SUMMARY:
The study aims to investigate the safety and tolerability of limb cryocompression in preventing of Chemotherapy-induced Peripheral Neuropathy via a newly developed limb cryocompression device in healthy subjects and cancer patients. The limb cryocompression device will be tested for its safety in delivering limb cryocompression and efficacy in improving the preservation of peripheral nerves during chemotherapy.

DETAILED DESCRIPTION:
The study consists of two parts. The first part of the study will consist of up to 18 healthy subjects to assess safety and tolerability of the new limb cryocompression device. The occurrence or lack of core hypothermia will be studied. The second part of the study will consist of 15 cancer patients recruited from the National University Hospital. Patients will undergo cryocompression over multiple cycles of chemotherapy to establish safety and tolerability of repeated therapy. Cryocompression of the limbs will be administered using cooling wraps attached to a cooling device. The limbs will be cooled from the digits to the elbow/knee.

ELIGIBILITY:
Inclusion Criteria:

1. For healthy subjects:

   * Age 21-80 years
   * Signed informed consent from patient or legal representative
   * No history of neuropathy
   * ECOG 0
   * No history of hospitalization in the past 6 months
2. For cancer patients:

   * Age 21- 80 years
   * Signed informed consent from patient or legal representative
   * Scheduled to receive weekly paclitaxel chemotherapy
   * Patients may receive other chemotherapy drugs alongside taxane e.g. Platinum/Herceptin.

Exclusion Criteria:

1. For healthy subjects:

   * Open skin wound or ulcers of the limbs
   * History of Raynaud's phenomenon, peripheral vascular disease, or poorly controlled diabetes
   * Pregnant women
2. For cancer patients:

   * Open skin wound or ulcers of the limbs
   * History of Raynaud's phenomenon, peripheral vascular disease, or poorly controlled diabetes
   * Pregnant women

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2021-11-03 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events in healthy volunteers, over the duration of a limb cryocompression cycle, as assessed by Common Terminology Criteria for Adverse Events 5.0 | During limb cryocompression procedure, 3 hours for healthy subject
  Defined as the number of subjects with treatment-related adverse events as assessed by CTCAE v5.0. Grade 1-5 refer to the severity of the adverse event with higher grade indicating greater severity. Grade 3 and above will be considered severe.
Difference in tolerance scores in healthy volunteers, over the duration of a limb cryocompression cycle, as assessed by Visual Analogue Scale for pain | During limb cryocompression procedure, 3 hours for healthy subject
  Defined as the number of subjects with treatment-related intolerance as assessed by tolerability scale, visual analog scale (VAS). On a scale of 0 to 10, a higher VAS score indicates higher intolerance. A score of 8 out of 10 will be considered dose-limiting intolerance.
Incidence of Treatment-Emergent Adverse Events in cancer patients, over the duration of a limb cryocompression cycle, as assessed by Common Terminology Criteria for Adverse Events 5.0 | During every cycle of paclitaxel chemotherapy (each cycle is 1 week) along with cryocompression which may last up to 4 hours, and for up to 12 cycles of weekly Paclitaxel treatment
  Defined as the number of patients with treatment-related intolerance as assessed by CTCAE v5.0. Grade 1-5 refer to the severity of the adverse event with higher grade indicating greater severity. Grade 3 and above will be considered severe.
Difference in tolerance scores in cancer patients, over the duration of a limb cryocompression cycle, as assessed by Visual Analogue Scale for pain | During every cycle of paclitaxel chemotherapy (each cycle is 1 week) along with cryocompression which may last up to 4 hours, and for up to 12 cycles of weekly Paclitaxel treatment
  Defined as the number of patients with treatment-related intolerance as assessed by tolerability scale, visual analog scale (VAS). On a scale of 0 to 10, a higher VAS score indicates higher intolerance. A score of 8 out of 10 will be considered dose-limiting intolerance.

SECONDARY OUTCOMES:
Difference in tolerance scores between various temperature and pressure using Common Terminology Criteria for Adverse Events 4.0 and Visual Analogue Scale for pain | During limb cryocompression procedure, 3 hours for healthy subject
  Difference in tolerance scores between various temperature and pressure as assessed by CTCAE v4.0 and tolerability scale, visual analog scale (VAS). On a scale of 0 to 10, a higher VAS score indicates higher intolerance. A score of 8 out of 10 will be considered dose-limiting intolerance.
Difference in qualitative symptom scores using the European Organisation of Research and Treatment of Cancer Quality of Life Questionnaire-CIPN twenty-item scale | Before start of weekly paclitaxel chemotherapy, at the end of 12 cycles of weekly paclitaxel treatment, at 3-, 6-, and 12-months post-treatment
  Difference in qualitative symptom scores using the EORTC QLQ-CIPN-20 scale before, at the end of paclitaxel chemotherapy with limb cryocompression, and at 3,6 and 12 months post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Raghav Sundar, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Loprinzi CL, Lacchetti C, Bleeker J, Cavaletti G, Chauhan C, Hertz DL, Kelley MR, Lavino A, Lustberg MB, Paice JA, Schneider BP, Lavoie Smith EM, Smith ML, Smith TJ, Wagner-Johnston N, Hershman DL. Prevention and Management of Chemotherapy-Induced Peripheral Neuropathy in Survivors of Adult Cancers: ASCO Guideline Update. J Clin Oncol. 2020 Oct 1;38(28):3325-3348. doi: 10.1200/JCO.20.01399. Epub 2020 Jul 14. PMID 32663120
- [Background] Windebank AJ, Grisold W. Chemotherapy-induced neuropathy. J Peripher Nerv Syst. 2008 Mar;13(1):27-46. doi: 10.1111/j.1529-8027.2008.00156.x. PMID 18346229
- [Background] Sundar R, Bandla A, Tan SS, Liao LD, Kumarakulasinghe NB, Jeyasekharan AD, Ow SG, Ho J, Tan DS, Lim JS, Vijayan J, Therimadasamy AK, Hairom Z, Ang E, Ang S, Thakor NV, Lee SC, Wilder-Smith EP. Limb Hypothermia for Preventing Paclitaxel-Induced Peripheral Neuropathy in Breast Cancer Patients: A Pilot Study. Front Oncol. 2017 Jan 10;6:274. doi: 10.3389/fonc.2016.00274. eCollection 2016. PMID 28119855
- [Background] Jordan B, Margulies A, Cardoso F, Cavaletti G, Haugnes HS, Jahn P, Le Rhun E, Preusser M, Scotte F, Taphoorn MJB, Jordan K; ESMO Guidelines Committee. Electronic address: clinicalguidelines@esmo.org; EONS Education Working Group. Electronic address: eons.secretariat@cancernurse.eu; EANO Guideline Committee. Electronic address: office@eano.eu. Systemic anticancer therapy-induced peripheral and central neurotoxicity: ESMO-EONS-EANO Clinical Practice Guidelines for diagnosis, prevention, treatment and follow-up. Ann Oncol. 2020 Oct;31(10):1306-1319. doi: 10.1016/j.annonc.2020.07.003. Epub 2020 Jul 30. No abstract available. PMID 32739407
- [Background] Bandla A, Tan S, Kumarakulasinghe NB, Huang Y, Ang S, Magarajah G, Hairom Z, Lim JSJ, Wong A, Chan G, Ngoi N, Ang E, Lee YM, Chan A, Lee SC, Thakor N, Wilder-Smith E, Sundar R. Safety and tolerability of cryocompression as a method of enhanced limb hypothermia to reduce taxane-induced peripheral neuropathy. Support Care Cancer. 2020 Aug;28(8):3691-3699. doi: 10.1007/s00520-019-05177-2. Epub 2019 Dec 6. PMID 31811482